CLINICAL TRIAL: NCT06544863
Title: Evaluation of Patient Care Support for Cirrhosis and/or Liver Transplants at Pitié Salpêtrière University Hospital
Brief Title: Evaluation of Patient Care Support for Cirrhosis and/or Liver Transplants
Acronym: PACCHUPS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231630
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis
Keywords: liver transplantation; alcohol; hepatitis B and C; metabolic syndrome
MeSH Terms: conditions — Fibrosis; Hepatitis B; Metabolic Syndrome | interventions — Data Collection; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis or suspected cirrhosis and/or TH patient: Patients with a diagnosis or suspected diagnosis of cirrhosis and/or TH managed at Pitié Salpêtrière University Hospital
  Interventions: Other: Data collection and blood sample

INTERVENTIONS:
Other: Data collection and blood sample — In addition to collecting medical data, additional blood samples will be collected in order to create a biological collection and identify biomarkers associated with the occurrence of cirrhosis-related complications, progression to TH and follow-up.

SUMMARY:
Cirrhosis is a major challenge in France, with a growing prevalence of 1,500 to 2,500 cases per million inhabitants, and the discovery of 150 to 200 new cases per million inhabitants each year. The main causes are alcohol, hepatitis B and C, and metabolic syndrome. Severe complications of cirrhosis, such as digestive hemorrhage, ascites, hepatic encephalopathy, infections and primary liver cancer, require frequent hospitalization and are more common in advanced stages of the disease. Around 15,000 deaths occur each year, affecting relatively young patients with an average age of 55. At the moment, the only treatment for these patients is liver transplantation (LT), although this is not feasible for all patients, and many complications may arise post LT.

Biological collections play an essential role in research, enabling the collection and storage of biological samples and clinical data to understand disease mechanisms and develop new therapeutic approaches or post-transplant follow-up. Longitudinal studies following the course of the disease offer a better understanding of risk factors and prognostic determinants. In this way, cirrhosis care support is constantly evolving, thanks to the evaluation of practices and the continuous improvement of patient care. For patients in whom TH is feasible, biological collections are also important for research and evaluation, and help improve post-TH care.

DETAILED DESCRIPTION:
Cirrhosis is a major challenge for healthcare professionals in France, with a growing prevalence in the country of over 1,500 to 2,500 diagnosed cases per million inhabitants, and the annual discovery of around 150 to 200 new cases per million inhabitants. The main causes of cirrhosis in France are excessive alcohol consumption, chronic viral hepatitis B and C, and metabolic syndrome. In the course of cirrhosis, severe complications can arise, such as digestive hemorrhage, ascites, hepatic encephalopathy, infections and primary liver cancer, requiring frequent hospitalization. These complications are more frequent in advanced cirrhosis, and may require liver transplantation. Around 15,000 deaths occur each year in France due to cirrhosis, affecting relatively young patients with an average age of 55. Currently, the only treatment for these patients is liver transplantation (LT), although this is not feasible for all patients, and many complications may arise post-LT. In order to improve the prognosis of patients with cirrhosis, several questions remain unanswered, such as the early diagnosis of cirrhosis in at-risk subjects, the identification of cirrhotic patients at high risk of complications, and the search for factors predictive of response to treatment of the various complications. The establishment of biological collections plays an essential role in research into cirrhosis and its complications, as well as the progression to TH and these complications. These biological collections enable the systematic collection and storage of biological samples and clinical data from cirrhosis and/or transplant patients. These resources are crucial for understanding the underlying mechanisms of the disease, identifying new diagnostic and prognostic biomarkers, and developing new therapeutic approaches.The development of a biological collection also offers the possibility of conducting longitudinal studies, tracking the progression of the disease in cirrhosis patients and/or post-TH. This enables a better understanding of risk factors, prognostic determinants and individual variations in disease progression. Thus, cirrhosis care support is constantly evolving, and the follow-up of a prospective cohort makes it possible to evaluate practices, determine prognostic factors and continually improve the management of patients, whether or not they are transplanted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients managed for cirrhosis or suspected cirrhosis and/or TH at Pitié Salpêtrière University Hospital
* Patients having been informed and having signed the consent to participate in the study.

Exclusion Criteria:

* Patient under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis or suspected diagnosis of cirrhosis and/or TH managed at Pitié Salpêtrière University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2040-03-19 (Estimated); Study Completion 2040-03-19 (Estimated)

PRIMARY OUTCOMES:
Evaluation of survival in cirrhosis and liver transplant patients. | During patient follow-up, for maximum 9 years
  Overall survival will be determined by the time between diagnosis and death of patients with cirrhosis or liver transplants.

SECONDARY OUTCOMES:
Assessment of the occurrence of complications (digestive hemorrhage, ascites, hepatic encephalopathy, infections and primary liver cancer) in patients with cirrhosis or liver transplants. | During patient follow-up, for maximum 9 years
  Patients will be followed longitudinally, and the occurrence and timing of complications (digestive bleeding, ascites, hepatic encephalopathy, infections and primary liver cancer) will be recorded for each patient.
Identification of clinico-biological predictors of cirrhosis-related or post-TH complications. | At inclusion
  Clinico-biological and imaging data collected from patients' diagnosis will be correlated with overall survival and the occurrence of complications (digestive hemorrhage, ascites, hepatic encephalopathy, infections and primary liver cancer).
Evaluation of the number of liver transplant patients with cirrhosis-related complications | During patient follow-up, for maximum 9 years
  The number of cirrhotic patients with complications (digestive hemorrhage, ascites, hepatic encephalopathy, infections and primary liver cancer) will then be followed longitudinally, and the number of patients requiring TH for these complications will be collected.
Determination of exosome profile in patients with tumor complication of cirrhosis or post-TH | During patient follow-up, for maximum 9 years
  Cirrhotic and TH patients will be followed longitudinally with regular sampling to monitor exosome profiles, sex steroid hormones and immune profiles (IFN-γ, TNF, IL10, IL12, TGF-β protein and transcriptomic profiles, etc.) during cirrhotic disease and TH (objectives 4, 5 and 6).
Determination of sex steroid hormone profile during cirrhotic disease or post-TH. | During patient follow-up, for maximum 9 years
  Cirrhotic and TH patients will be followed longitudinally with regular sampling to monitor exosome profiles, sex steroid hormones and immune profiles (IFN-γ, TNF, IL10, IL12, TGF-β protein and transcriptomic profiles, etc.) during cirrhotic disease and TH (objectives 4, 5 and 6).
Immune status in cirrhotic or post-TH patients (IFN-γ, TNF, IL10, IL12, TGF-β protein and transcriptome profiles ...) | During patient follow-up, for maximum 9 years
  Cirrhotic and TH patients will be followed longitudinally with regular sampling to monitor exosome profiles, sex steroid hormones and immune profiles (IFN-γ, TNF, IL10, IL12, TGF-β protein and transcriptomic profiles, etc.) during cirrhotic disease and TH (objectives 4, 5 and 6).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Digestive Surgery Department, Pitié-Salpêtrière Hospital, Paris
  - Intensive Care Unit, Pitié Salpêtrière Hospital, Paris
  - Pitié Salpêtrière University Hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.